CLINICAL TRIAL: NCT00724984
Title: Phase I/II Dose-Escalation Study of the Pan-Histone Deacetylase (HDAC) Inhibitor PCI-24781 in Lymphoma
Brief Title: Study of the Safety and Tolerability of PCI-24781 in Patients With Lymphoma
Acronym: PCYC-0403
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0403
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin
Keywords: PCI-24781; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle Cell; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral | interventions — abexinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PCI-24781

INTERVENTIONS:
Drug: PCI-24781 — Phase I Dose Escalation: Up to 5 cohorts will receive PCI-24781 orally at doses starting at 30mg/m2 two times a day approximately 4-6 hours apart ("BID"), up to 90mg/m2 administered 5 days/week during the first 21 days of each 28 day cycle until the maximum tolerated dose (MTD) is reached. If a dose limiting toxicity (DLT) occurs, then the next cohort will receive PCI-24781 BID for 7 days every other week (2 times in a 28 day cycle).
  Phase II Efficacy Evaluation: All patients will receive PCI-24781 orally at the dosage and regimen determined in Phase I.

SUMMARY:
The first part of the study will determine the highest dose of study drug that can be taken without causing serious side effects in patients with lymphoma. The appropriate dose determined from the first part of the study will be used in the second part of the study to assess disease response in 2 different types of lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* • age ≥ 18 years

  * Phase I: Any measurable, histologically confirmed, and previously treated lymphoma
  * Phase II: Measurable, histologically confirmed, and previously treated lymphoma in one of the following categories:

    1. Follicular non-Hodgkin's Lymphoma
    2. Mantle cell lymphoma
  * Ability to swallow oral capsules without difficulty
  * Estimated life expectancy > 12 weeks
  * ECOG performance status ≤ 1
  * Willing and able to sign a written informed consent

Exclusion Criteria:

* • More than four prior systemic treatment regimens (not counting maintenance rituximab; salvage therapy/conditioning regimen preceding autologous bone marrow transplantation [ABMT] and ABMT count as one regimen)

  * Allogeneic bone marrow transplant
  * Immunotherapy, chemotherapy, radiotherapy or experimental therapy within 4 weeks before first day of study drug dosing
  * Major surgery within 4 weeks before first day of study drug dosing
  * CNS lymphoma or a history of meningeal carcinomatosis
  * Prior treatment with an HDAC inhibitor (unless for treatment of Mycosis fungoides or Sézary syndrome)
  * Creatinine > 1.5 x institutional upper limit of normal (ULN) or creatinine clearance ≤ 50 mL/min
  * Total bilirubin > 1.5 x institutional ULN (unless elevated from documented Gilbert's syndrome)
  * AST and ALT > 2.5 x institutional ULN
  * Platelet count < 75,000/µL for Phase I and <100,000>µL for Phase II
  * Absolute neutrophil count (ANC) < 1500/µL
  * Malabsorption
  * Corticosteroids > 20 mg prednisone equivalent per day (topical, inhaled, or nasal corticosteroids are permitted)
  * Concurrent therapeutic anticoagulation (Phase I only)
  * Uncontrolled illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements
  * Risk factors for, or use of drugs known to prolong QTc interval or that may be associated
  * QTc prolongation (defined as a QTc ≥ 450 msecs) or other significant ECG abnormalities including 2nd degree AV block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min). If the screening ECG has a QTc ≥ 450 msecs, the ECG can be submitted for a centralized, cardiologic evaluation.
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within the past 6 months.
  * For patients with history of myocardial infarction, congestive heart failure, abnormal left ventricular ejection fraction (LVEF), and/or prior anthracycline exposure, LVEF < 50%, as assessed by ventriculography (nuclear or heart catheterization) or echocardiogram, when performed within 28 days of first dose of study drug.
  * For patients with history of coronary artery disease, a cardiac stress test (either exercise or pharmacologic) that demonstrates clinically significant abnormalities when performed within 28 days of first dose of study drug.
  * Known HIV infection.
  * Other medical or psychiatric illness or organ dysfunction which, in the opinion of the investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of the study agent.
  * Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound).
  * Women of child-bearing potential, or sexually active men, unwilling to use adequate contraceptive protection during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Graef, MD, Study Director — Pharmacyclics LLC.
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Northwestern University Medical School, Chicago, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Vermont and Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Result] Buggy JJ, Cao ZA, Bass KE, Verner E, Balasubramanian S, Liu L, Schultz BE, Young PR, Dalrymple SA. CRA-024781: a novel synthetic inhibitor of histone deacetylase enzymes with antitumor activity in vitro and in vivo. Mol Cancer Ther. 2006 May;5(5):1309-17. doi: 10.1158/1535-7163.MCT-05-0442. PMID 16731764
- See also: Related Info — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1(30mg/m2,5days/wk)/Phase 1 | Cohort 2(45mg/m2,5days/wk)/Phase 1 | Cohort 3(45mg/m2,7days/wk)/Phase 1 | Cohort 4(60mg/m2,7days/wk)/Phase 1 | Follicular/Phase II | Mantle Cell Lymphoma/Phase II
Started | 5 | 8 | 3 | 9 | 16 | 14
Completed | 4 | 7 | 3 | 7 | 12 | 9
Not Completed | 1 | 1 | 0 | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1(30 mg/m2, 5days/wk)/Phase 1 | Cohort 2(45 mg/m2, 5days/wk)/Phase 1 | Cohort 3(45 mg/m2, 7days/wk)/Phase 1 | Cohort 4(60 mg/m2,7days/wk)/Phase 1 | Follicular/Phase II | Mantle Cell Lymphoma/Phase II | Total
Number analyzed (Participants) | 5 | 8 | 3 | 9 | 16 | 14 | 55
Age, Continuous [Median (Full Range); unit: years] | 68 [40 to 75] | 67 [47 to 76] | 62 [32 to 79] | 66 [44 to 76] | 62 [36 to 81] | 67 [59 to 77] | 66 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 3 | 8 | 12 | 30
  Male | 4 | 3 | 2 | 6 | 8 | 2 | 25
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 3 | 9 | 16 | 14 | 55

OUTCOME MEASURES:

1. Primary Outcome: Phase I (Dose Escalation Phase): MTD and DLTs of PCI-24781 Administered Twice Daily (BID) Measure: Disease Response
Description: Number of patients experienced DLT in each cohort
Time Frame: From the Date of PCI-24781 first administration to Cycle 2 Day 1
Measure: Number; unit: participants
Arm/Group | Cohort 1(30 mg/m2, BID, 5days/wk)/Phase I | Cohort 2(45 mg/m2, BID, 5days/wk)/Phase I | Cohort 3(45 mg/m2, BID, 7days/wk)/Phase I | Cohort 4(60 mg/m2, BID, 7days/wk)/Phase I
Number analyzed (Participants) | 3 | 7 | 3 | 8
participants | 0 | 3 | 0 | 2

2. Primary Outcome: Phase II: Overall Response Rate (CR+PR)
Time Frame: From first response assessment (day 22 to 28 of Cycle 2) to last response assessment on day 22-28 in even-numbered cycles
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Follicular/Phase II (Efficacy) | Mantle Cell Lymphoma/Phase II (Efficacy)
Number analyzed (Participants) | 16 | 14
Percentage of Participants | 56.3 [29.9 to 80.2] | 21.4 [4.66 to 50.8]

ADVERSE EVENTS:
Arm/Group | Cohort 1(30 mg/m2, 5days/wk)/Phase I | Cohort 2(45 mg/m2, 5days/wk)/Phase I | Cohort 3(45 mg/m2, 7days/wk)/Phase I | Cohort 4(60 mg/m2,7days/wk)/Phase I | Follicular/Phase II | Mantle Cell Lymphoma/Phase II
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/8 | 0/3 | 3/9 | 6/16 | 5/14
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 3/3 | 9/9 | 16/16 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1(30 mg/m2, 5days/wk)/Phase I (N=5) | Cohort 2(45 mg/m2, 5days/wk)/Phase I (N=8) | Cohort 3(45 mg/m2, 7days/wk)/Phase I (N=3) | Cohort 4(60 mg/m2,7days/wk)/Phase I (N=9) | Follicular/Phase II (N=16) | Mantle Cell Lymphoma/Phase II (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
ANAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
ENCEPHALITIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
ANURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1(30 mg/m2, 5days/wk)/Phase I (N=5) | Cohort 2(45 mg/m2, 5days/wk)/Phase I (N=8) | Cohort 3(45 mg/m2, 7days/wk)/Phase I (N=3) | Cohort 4(60 mg/m2,7days/wk)/Phase I (N=9) | Follicular/Phase II (N=16) | Mantle Cell Lymphoma/Phase II (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 4 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 4 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 4 | 0 | 2 | 10 | 4
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
EYE SWELLING (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
EYELID IRRITATION (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
MIOSIS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 3 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 7 | 3
DIARRHOEA (Gastrointestinal disorders) | 0 | 3 | 0 | 5 | 8 | 7
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 1
ERUCTATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 2
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 4 | 1
GLOSSODYNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 11 | 7
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
RETCHING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 7 | 3
CHEST DISCOMFORT (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
CHILLS (General disorders) | 0 | 1 | 0 | 1 | 1 | 5
EARLY SATIETY (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
FATIGUE (General disorders) | 4 | 6 | 1 | 2 | 10 | 8
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
LOCALISED OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0 | 1 | 2 | 5
PAIN (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
PYREXIA (General disorders) | 1 | 1 | 0 | 0 | 3 | 1
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0
CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
INFECTED BITES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 4
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 2 | 0 | 3 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM ST-T CHANGE (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
HAEMOGLOBIN (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
HEART RATE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
TROPONIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 4 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 3 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 2
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
CLUBBING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
AREFLEXIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
ATAXIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 3 | 0 | 2 | 3 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 3
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 1 | 5 | 3
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPOGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
INTENTION TREMOR (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MOTOR DYSFUNCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
PAROSMIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 6 | 7
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2 | 1 | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OBLITERATIVE BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
RALES (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
RESPIRATORY TRACT OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 2 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
SKIN BURNING SENSATION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL COLDNESS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No